CLINICAL TRIAL: NCT00638287
Title: Inter-Assay Growth Hormone and IGF-I Variability
Status: Withdrawn | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Inter-Assay Growth Hormone and IGF-I Variability, CSMC
Other Study IDs: 10638
Record Dates: First submitted 2008-01-11; First posted 2008-03-19 (Estimated); Last update posted 2008-10-06 (Estimated); Status verified 2008-09

CONDITIONS: Acromegaly; Growth Hormone Deficiency
Keywords: Subjects with pituitary disease undergoing testing for GH; deficiency; Subjects with suspicion for (or diagnosis of) acromegaly; undergoing OGTT testing; Normal controls without evidence of pituitary dysfunction
MeSH Terms: conditions — Acromegaly; Dwarfism, Pituitary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Group I Growth Hormone Deficiency (GHD): subjects with pituitary disease undergoing testing for GH deficiency: GHRH-ARG Test, collect total of 84 cc whole blood.
  2. Group II Acromegaly: subjects with suspicion for (or diagnosis of) acromegaly undergoing OGTT Test, collect total of 48 cc whole blood.
  3. Group III Normal Controls: subjects without evidence of pituitary dysfunction undergoing OGTT Test, collect total of 136 cc whole blood.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to demonstrate the degree of variability in commercially available assays for Growth Hormone measurement in the context of clinical decision making for Growth Hormone (GH) deficiency and Acromegaly and to determine variability among IGF-I inter-assay samples obtained at the time of Growth-Hormone Releasing Hormone Arginine Testing and Oral Glucose Tolerance Testing.

DETAILED DESCRIPTION:
This research will explore the variability of GH and IGF-1 measurements by commercially available tests. The hypothesis is that the variability in GH and IGF-1 measurement will be sizable enough that different conclusions would be drawn in patient case decision making in the diagnosis and management of GH deficiency and acromegaly.

In order to correctly diagnose disorders of growth hormone secretion, either deficiency or excess, it is necessary to have the accurate measurement of GH (growth hormone) serum and Insulin-like growth factor (IGF-1).

For this study, subjects will be asked to give the Investigators additional blood during either an OGTT (a test for acromegaly) or a growth hormone stimulation test (GHRH-arginine stimulation). Ordinarily, blood would be measured at the beginning and end of the OGTT, and for the GHRH-arginine it would be measured one half hour before the test and then every half hour for 2 hours.

For this study, subjects will provide us with additional blood at the times when blood is drawn for the clinically-indicated tests. No additional needle sticks will be necessary and taking the additional blood will not interfere with the clinical test.

The test we will be doing with the additional blood will be identical to the tests we ordinarily do, but will be done by a different lab. We are testing to see if these results would be the same as our usual lab.

The study population will include 1) subjects with pituitary disease undergoing testing for GH deficiency (GHRH arginine stimulation test), 2) subjects with suspicion of acromegaly undergoing the oral glucose tolerance test (oGTT), and 3) normal controls undergoing both the GHRH Arginine test and the oGTT. Patients from all groups will have their blood drawn for the measurement of IGF-1. The serum from each test will be aliquoted and sent to the designated labs.

For subject groups 1 and 2, this study poses no more than minimal risk, as it involves procedures that do not go beyond clinical care. For healthy controls, we know that participants will be asked to undergo testing that would not normally be required, and therefore feel that the study poses more than minimal risk.

For the primary endpoint research samples will be compared to samples sent to the usual clinical lab, and diagnoses made based on research samples will be compared to clinical samples.

For secondary endpoints, each result from a commercially available assay will be correlated to another corresponding method of analysis of the same hormone from the same time point by using the Bland-Altman analysis wherein the difference between two methods is compared to the mean of the two methods. Each sample will be compared to the sample used for clinical evaluation.

Information from the medical records will be obtained and correlated with the lab test results.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female age 18+
2. Clinical indication for testing GH response to secretagogue testing to evaluate for GHD OR clinical indication for testing for GH response to oral glucose load (75grams of glucose) to evaluate for Acromegaly either for diagnosis OR normal volunteer for control group.

   * Normal volunteers will be screened for evidence of pituitary endocrine dysfunction prior to Oral Glucose Tolerance Testing (OGTT) and Growth Hormone Releasing Hormone - Arginine Testing (GHRH-ARG).
3. Able to provide informed consent

Exclusion Criteria:

1. Subjects taking GH
2. Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: tertiary referral center
Sampling Method: Probability Sample
Enrollment: 171 (Estimated)
Dates: Start 2007-11; Study Completion 2011-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John Carmichael, MD, Principal Investigator — Cedars-Sinai Medical Center